CLINICAL TRIAL: NCT03355885
Title: Impact of Early Diagnosis Algorithm for Early-onset Pneumonia Diagnosis on Prognosis of Patients With Out-of-hospital Cardiac Arrest
Brief Title: Early-onset Pneumonia After Out-of-hospital Cardiac Arrest
Acronym: PP-ACR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PP-ACR
Record Dates: First submitted 2017-11-23; First posted 2017-11-28 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-10

CONDITIONS: Out-of-Hospital Cardiac Arrest
Keywords: early onset pneumonia; out-of-hospital cardiac arrest; prognosis; antibiotic
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Early-onset pneumonia after out-of-hospital cardiac arrest is frequent. An association between early-onset pneumonia and an increase in morbidity has been reported in this population. The diagnosis of early-onset pneumonia inpatients with out-of-hospital cardiac arrest may be challenging as diagnosis criteria are unspecific in this setting. On the other hand some studies have reported an association between early antibiotics and better prognosis in patients with out-of-hospital cardiac arrest suggesting that early diagnosis and treatment of pneumonia would benefit to patients. Nonetheless, adminitration of antibiotics to any patients with out-of-hospital cardiac arrest would expose to antibiotic patients without infection and woould participate to increase in antibiotic resistance.

Therefore, the PP-ACR study aims to evaluate the impact of a diagnosis algorithm including blinded sampling protected brushes on early-onset pneumonia treatment and patient prognosis after out-of-hospital cardiac arrest.

DETAILED DESCRIPTION:
This study is a single centre observational study with a before - after design.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted for out-of-hospital cardiac arrest and treated with hypothermia

Exclusion Criteria:

* age less than 18
* consent withdrawal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted for out-of-hospital cardiac arrest in intensive care who and treated with hypothermia
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2016-10-03 (Actual); Primary Completion 2018-05-31 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
delay between intensive care admission and antibiotic initiation | first 5 days
delta respiratory SOFA score between Day 1 and day 3 | first 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lemee P, Chapalain X, Bailly P, Sparrow RL, Jean-Michel V, Prat G, Renault A, Tonnelier JM, Aubron C. PROACTIVE SCREENING ALGORITHM FOR EARLY-ONSET PNEUMONIA IN PATIENTS WITH OUT-OF-HOSPITAL CARDIAC ARREST: A BEFORE-AFTER IMPLEMENTATION STUDY. Shock. 2024 Jul 1;62(1):13-19. doi: 10.1097/SHK.0000000000002347. Epub 2024 Mar 25. PMID 38661180